CLINICAL TRIAL: NCT04505683
Title: A Phase 2, Randomized, Double-blind, Positive-control, Multicenter, Prospective Study to Assess Efficacy and Safety of Intravenous Benapenem in Patients With Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)
Brief Title: A Study to Assess Efficacy and Safety Intravenous Benapenem in Patients With Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5081-II-2001
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Complicated Urinary Tract Infection Including Acute Pyelonephritis
MeSH Terms: interventions — benapenem; Ertapenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test drug arm (Experimental): Benapenem for IV injection administered as a 1-gram IV infusion over 30 min once daily for 7 to 14 days.
  Interventions: Drug: Benapenem
- active control arm (Active Comparator): Ertapenem for IV injection administered as a 1-gram IV infusion over 30 min once daily for 7 to 14 days.
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Benapenem — Benapenem for IV injection administered as a 1-gram IV infusion
  Arms: test drug arm
Drug: Ertapenem — Ertapenem for IV injection administered as a 1-gram IV infusion
  Arms: active control arm

SUMMARY:
A Study to Assess Efficacy and Safety Intravenous Benapenem in Patients With Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-75 years
2. Have a diagnosis of cUTI or AP as defined below:

   1. cUTI definition:

      * At least Two of the following signs and symptoms:

        * Chills, rigors, or fever; fever must be observed and documented by a health care provider (tympanic temperature ≥37.3°C)
        * Flank pain or Lower abdominal pain
        * Dysuria, urgency to void, or increased urinary frequency
        * Nausea or vomiting
        * Costovertebral angle tenderness or renal percussive pain on physical examination.
        * Blood leukocytes above upper limit of normal value

      And at least One of the following risk factors for cUTI:
      * Implanted urinary tract instrumentation (e.g., nephrostomy tube, ureteric stents), ongoing intermittent bladder catheterization, or presence of an indwelling bladder catheter (Note: bladder catheters prior to Screening should be expected to remove during study period
      * post-void residual urine volume of ≥ 100 mL;
      * Obstructive uropathy (e.g. bladder outlet obstruction, nephrolithiasis, prostatic hyperplasia) that is expected to be removed during study drug therapy;
      * Perioperative urinary tract infection.
   2. AP definition: And at least One of the following signs and symptoms:

      * Chills, rigors, or fever; fever must be observed and documented by a health care provider (tympanic temperature ≥37.3°C）；
      * Flank pain
      * Dysuria, urgency to void, or increased urinary frequency
      * Nausea or vomiting
      * Costovertebral angle tenderness or renal percussive pain on physical examination.
      * Blood leukocytes above upper limit of normal value
3. Patients or legal representatives can be able to provide informed consent

Exclusion Criteria:

1. Receipt of potentially effective antibiotic therapy more than 24h within 72 h prior to randomization
2. Anticipated concomitant use of other systemic antibiotic drugs during the study period
3. Anticipated continnue to preventive anti-infectious therapy after cUTI patients completed investigational drug treatment
4. Presence of any known or suspected disease or condition as following:

   * Uncomplicated urinary tract infection (uUTI)
   * Fungal Urinary tract infection
   * Perinephric or renal corticomedullary abscess
   * Polycystic kidney disease
   * Urinary tuberculosis
   * Obstructive uropathy(e.g.congenital malformation) unable to remove during treatment.
   * Ideal loop surgery or vesicoureteral reflux
   * Permannent bladder catheterization or long term indwelling nephrostomy tube
   * Previous or planned renal transplantation
   * Patients undergoing dialysis"
5. Confirmed or suspected acute or chronic bacterial prostatitis, orchitis, or epididymitis
6. Confirmed or suspected sexually transmitted disease,e.g. gonorrhea and syphilis
7. Confirmed or suspected non-renal source of infection (e.g., infective endocarditis, osteomyelitis, meningitis, pneumonia)
8. Trauma to the pelvis or urinary tract within 7days before enrollment
9. Rapid onset or life-threatening diseases, such as septic shock, respiratory failure, sepsis, etc;
10. Severe cardiovascular and cerebrovascular diseases, acute myocardial infarction, acute ischemic stroke, acute Hemorrhagic stroke or intravascular intervention within recently 3 months
11. Known or suspected central nerve system disorders, prone to epilepsy(e.g severe carebral arteriosclerosis)
12. Known history of immunodeficiency diease, e.g.AIDS or human immunodeficiency virus (HIV) infection,hematologic malignancy, bone marrow transplant, or receiving immunosuppressive therapy such as cancer chemotherapy, medications for the rejection of transplantation, and long term use of systemic corticosteroids;
13. Use of valproic acid or probenecid within 30 days before enrollment or during study period.
14. Hepatic impairment at Screening, evidenced as:

    * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3x upper limit of normal (ULN);
    * total bilirubin >1.5x ULN;
    * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2x upper limit of normal (ULN) and total bilirubin > ULN; Creatinine clearance (CrCl) of <60 mL/min, as estimated by the Cockcroft-Gault formula: estimated Creatinine Clearance (eC_Cr) [mL/min]=((140-Age [yrs]) × Body Weight [kg] × [0.85 if Female])/(72 × Serum Creatinine [mg⁄dL])
15. Known allergic to β-lactam drugs or in an allergic state
16. Confirmed or suspected alcohol or drug abuse history
17. Patients with other mental disorders who are unable or unwilling to cooperate.
18. Pregnant or breastfeeding women or plan to pregnant and unwilling to take contraceptive methods
19. Participants in other clinical trials within 3 months before enrollment.
20. Other situations that the investigators considers not suitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with clinical cure at test-of-cure (TOC) visit | Day 7 +/- 1 days after the end of treatment
  Clinical cure is defined as complete resolution of signs,symptoms and related laboratory tests of cUTI or AP that were present at baseline and no new symptoms, such that no further antimicrobial therapy is warranted.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China